CLINICAL TRIAL: NCT01263249
Title: Continuous Femoral Nerve Blocks: Effects of Catheter Tip Location Relative to the Femoral Nerve on Sensory and Motor Function
Brief Title: Effects of Catheter Tip Location Relative to the Femoral Nerve on Sensory and Motor Function
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Brian Ilfeld, M.D., M.S., University of California, San Diego, Department of Anesthesiology
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Volunteer Anterior Posterior
Record Dates: First submitted 2010-12-16; First posted 2010-12-20 (Estimated); Last update posted 2011-06-14 (Estimated); Status verified 2011-06

CONDITIONS: Continuous Femoral Nerve Blocks in Healthy Volunteers
Keywords: Femoral; Nerve Block; Anterior; Posterior; Continuous Infusion; Perineural Catheter; Volunteer; Lower Extremity Nerve Blocks

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Catheter Anterior to Femoral Nerve (Active Comparator): Each subject will have one lower extremity (Right or Left) randomized to receive a perinural catheter, placed anterior to the femoral nerve, with a continuous infusion of local anesthetic and then the outcomes will be measured.
  Interventions: Procedure: Catheter Anterior to the Femoral Nerve
- Catheter Posterior to Femoral Nerve (Active Comparator): Each subject will have the opposite lower extremity (Right or Left) randomized to receive a perinural catheter, placed posterior to the femoral nerve, with a continuous infusion of local anesthetic and then the outcomes will be measured.
  Interventions: Procedure: Catheter Posterior to the Femoral Nerve

INTERVENTIONS:
Procedure: Catheter Anterior to the Femoral Nerve — Extremity randomized to Anterior Placement will be given a peripheral nerve block with the catheter placed just anterior to the femoral nerve. 4cc of Ropivicaine will be administered continuously every hour by a pain pain pump and the outcome measures will be tested.
  Arms: Catheter Anterior to Femoral Nerve
Procedure: Catheter Posterior to the Femoral Nerve — Extremity randomized to Posterior Placement will be given a peripheral nerve block with the catheter placed just posterior to the femoral nerve. 4cc of Ropivicaine will be administered continuously every hour by a pain pain pump and the outcome measures will be tested.
  Arms: Catheter Posterior to Femoral Nerve

SUMMARY:
To determine if the way local anesthetic, or numbing medication, is delivered through a tiny tube next to the nerves that go to the thigh affects the strength and sensation in the thigh.

DETAILED DESCRIPTION:
Specific Aim: Research study to test the hypothesis that differing the location of the perineural catheter tip during a continuous femoral nerve block (anterior vs. posterior) impacts quadriceps muscle strength. These results will help define the optimal perineural catheter tip location relative to the femoral nerve used for continuous peripheral nerve blocks and help guide both clinical care and future research in this clinically-relevant area.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or over
* Willing to have bilateral femoral perineural catheters placed with a subsequent ropivacaine infusion and motor/sensory testing for 6 hours, requiring an overnight stay in the UCSD GCRC/CTRI to allow dissipation of local anesthetic infusion effects by the following morning

Exclusion Criteria:

* current daily analgesic use
* opioid use within the previous 4 weeks
* any neuro-muscular deficit of either femoral nerves and/or quadriceps muscles
* body mass index > 30 kg/m2
* pregnancy
* incarceration

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Estimated)
Dates: Start 2010-01; Primary Completion 2011-04 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Quadriceps femoris muscle strength | percentage of baseline muscle strength six hours after infusion initiation
  The primary end point will be the quadriceps femoris maximum voluntary isometric contraction (MVIC) expressed as a percentage of the pre-ropivacaine MVIC: post / pre x 100; with the two sides of each subject compared with each other

CONTACTS AND LOCATIONS:
Overall Officials: Brian M Ilfeld, M.D., M.S., Principal Investigator — University of California, San Diego
Locations (1):
- UCSD Medical Center, Hillcrest, San Diego, California, United States